CLINICAL TRIAL: NCT02059356
Title: Prevalence of High Ammonia Levels in Patients With Cognitive Impairment. Does Treatment Help?
Brief Title: Ammonia Levels and Cognitive Impairment
Status: Terminated | Type: Observational
Why Stopped: Low patient recruitment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00048143
Record Dates: First submitted 2014-01-06; First posted 2014-02-11 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Dementia; Cognitive Decline; Cognitive Impairment; Developmental Delay
Keywords: Dementia; Alzheimer's; Alzheimers; Cognitive decline; Cognitive impairment; Memory loss; Memory disorder; Forgetfulness; Confusion; Senile; Demented; Developmental delay; Portal systemic shunting; High ammonia level; Elevated ammonia level
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Learning Disabilities; Memory Disorders; Confusion; Hyperammonemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-cirrhotic patients with cognitive impairment

SUMMARY:
The purpose and objective of this study is to determine the prevalence of elevated ammonia levels in subjects with cognitive impairment, and to observe if treating the cause of the elevated ammonia level improves mental status. This study does not include any imaging, treatment,or interventions, other than the blood draws. The blood draws will be taken to assess blood ammonia level and liver function. If the the ammonia level is not elevated, no further lab draws will occur. If the ammonia level is elevated, liver function is normal, and a cause for the high ammonia level is revealed with a plan for clinical treatment by the subjects' physician, then two more blood draws will occur; one prior to treatment, and one 3 months after treatment. The main risk to subjects is related to the blood draw (i.e. momentary discomfort, bruising, infection, bleeding, clotting or fainting), and there is a potential loss of confidentiality. A paired student t test will be done with the two later blood to compare objective data.

ELIGIBILITY:
Inclusion Criteria:

* cognitive decline (suspected or documented)
* able to get blood drawn

Exclusion Criteria:

* liver disease/cirrhosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of assisted living center or the general public
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in blood ammonia level | Baseline, Pretreatment and 3 months after treatment

SECONDARY OUTCOMES:
Change in mini-status examination | Prior to treatment and 3 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States